CLINICAL TRIAL: NCT04758078
Title: Inhaled Budesonide in Transient Tachypnea of the Newborn: A Randomized, Placebo-controlled Study
Brief Title: Inhaled Budesonide in Transient Tachypnea of the Newborn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Sirin Mneimneh, Pediatrician, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 09102020
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Distress
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroids (Experimental): Patients will receive inhaled corticosteroids (Budesonide 2 mL = 1000 microgram)
  Interventions: Other: Inhaled corticosteroids
- Placebo (Placebo Comparator): Patients will receive nebulized 0.9% saline
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Inhaled corticosteroids — Budesonide 2 mL = 1000 microgram will be given within 6 hours of birth and the second dose will be given after 12 hours
  Arms: Corticosteroids
Other: Placebo — Nebulized 0.9% saline will be given four times per day
  Arms: Placebo

SUMMARY:
Background: Transient tachypnea of the newborn (TTN) caused by lung edema resulting from delayed absorption of fetal alveolar lung fluid and is a common cause of admission of late preterm and full-term infants to neonatal intensive care units. Infant born by C-section and those with perinatal asphyxia, umbilical cord prolapse or certain maternal condition (asthma, diabetes, or analgesia) are more prone to develop TTN. Conventional treatment involves appropriate oxygen administration and continuous positive airway pressure in some cases. Hastening the clearance of lung liquid should shorten the duration of the symptoms and reduce complications.

Objectives: This study aims to determine the effectiveness of inhaled budesonide in the treatment of this disorder through determining whether it reduces the duration of oxygen therapy and respiratory symptoms and shortens hospital stay in term infants with transient tachypnea of the newborn

ELIGIBILITY:
Inclusion Criteria:

* Late preterm and term infants (post-menstrual age ≥ 34 weeks) delivered by Cesarean section or vaginal delivery
* Diagnosis of transient tachypnea of the newborn
* The need for Continuous positive airway pressure (CPAP) >6 hours to obtain the oxygen saturation >92%

Exclusion Criteria:

* Meconium aspiration syndrome;
* Respiratory distress syndrome
* Congenital heart Disease
* Non respiratory disorders causing tachypnea (polycythemia or hypoglycemia) resolving with treatment of the disorder
* Pneumonia by chest x-ray
* Suspected sepsis/bacteremia
* Prenatal steroids

Min Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of respiratory distress | within 48 hours
  Transient tachypnea of the newborn clinical score

SECONDARY OUTCOMES:
Assessment of time to spontaneous breathing | with 48 hours
  Time to spontaneous unsupported breathing of room air (in hours)

CONTACTS AND LOCATIONS:
Overall Officials: Sirin Mneimneh, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon